CLINICAL TRIAL: NCT02017106
Title: Randomized Clinical Trial of Concomitant or Sequential Phlebectomy After Endovenous Laser Therapy for Varicose Veins
Brief Title: Concomitant or Sequential Phlebectomy After Endovenous Laser Therapy for Varicose Veins
Acronym: EVLTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVLTAP
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Varicose Veins; Endovenous Laser Ablation; Phlebectomies
Keywords: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concomitant phlebectomies (Experimental): Removal of varicose tributaries during Endovenous laser ablation
  Interventions: Procedure: Endovenous Laser ablation and concomitant phlebectomies; Procedure: Endovenous Laser ablation and sequential phlebectomies
- Sequential Phlebectomies (Active Comparator): Endovenous laser ablation only
  Interventions: Procedure: Endovenous Laser ablation and concomitant phlebectomies; Procedure: Endovenous Laser ablation and sequential phlebectomies

INTERVENTIONS:
Procedure: Endovenous Laser ablation and concomitant phlebectomies
Procedure: Endovenous Laser ablation and sequential phlebectomies

SUMMARY:
Varicose veins of the leg often have superficial tributaries, which are often symptomatic and a major reason for coming to the doctor. When treating the main varicose vein inside the leg, some doctors prefer to remove these tributaries while others prefer to leave them. This trial aims to see if it is better to remove these veins at the time of the first laser procedure or better to leave them and only remove them when asked.

DETAILED DESCRIPTION:
Endovenous laser therapy (EVLT) for varicose veins is associated with high initial occlusion rates, minimal complications and low recurrence rates at 5 years. Randomized trials and meta-analyses have confirmed the efficacy of EVLT in comparison with surgery and other endovenous techniques. There is also evidence that it may be associated with early quality of life (QoL) benefits compared with surgery. The general efficacy of EVLT has therefore been demonstrated and current research focuses on refinement of the procedure. A fundamental question concerns the management of residual varicosities following truncal laser ablation. One approach is to leave these varicosities to regress untouched, minimizing the procedure time and surgical trauma6. This approach, however, is associated with a significant number of secondary and tertiary interventions (sclerotherapy and/or ambulatory phlebectomy). Another option is to combine in a single procedure ambulatory phlebectomy with initial truncal laser ablation (EVLTAP). The aim of this randomized controlled trial was to assess the advantages of performing ambulatory phlebectomy as a concomitant procedure to truncal laser ablation.

ELIGIBILITY:
Inclusion Criteria:

* primary, symptomatic, unilateral varicose great saphenous veins (GSV), with isolated saphenofemoral junction (SFJ) incompetence and GSV reflux on venous duplex imaging,
* perigenicular vein diameter exceeding 4 mm,
* acceptance by the patient of a local anaesthetic procedure.

Exclusion Criteria:

* saphenopopliteal, small saphenous or deep venous incompetence on duplex imaging
* did not give consent to trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Disease specific QoL (AVVQ) | 5 years

SECONDARY OUTCOMES:
Number of secondary procedures | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hull Royal Infirmary, Hull, Humberside, United Kingdom

REFERENCES:
- [Result] Carradice D, Mekako AI, Hatfield J, Chetter IC. Randomized clinical trial of concomitant or sequential phlebectomy after endovenous laser therapy for varicose veins. Br J Surg. 2009 Apr;96(4):369-75. doi: 10.1002/bjs.6556. PMID 19283745